CLINICAL TRIAL: NCT01121016
Title: Randomized Double-blind Placebo-controlled Study of add-on Montelukast to Inhaled Budesonide in the Treatment of Nonasthmatic Eosinophilic Bronchitis
Brief Title: Efficacy and Safety of add-on Montelukast to Inhaled Budesonide in the Treatment of Nonasthmatic Eosinophilic Bronchitis
Acronym: NAEB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Chuang Cai/ Associate Professor, Guangzhou Institute of Respiratory Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: moneb
Record Dates: First submitted 2010-05-11; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2009-09

CONDITIONS: Nonasthmatic Eosinophilic Bronchitis
Keywords: NAEB, chronic cough, montelukast, induced sputum
MeSH Terms: conditions — Chronic Cough | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination therapy (Active Comparator): combination therapy with inhaled budesonide and oral montelukast
  Interventions: Drug: Montelukast
- monotherapy (Placebo Comparator): monotherapy with inhaled budesonide and placebo of montelukast
  Interventions: Other: placebo to montelukast

INTERVENTIONS:
Drug: Montelukast — 10mg, qn, 4 weeks
  Other Names: Singulair
  Arms: combination therapy
Other: placebo to montelukast — same appearance, flavor, weight, and size to montelukast pills, 1 pill daily, for 4 weeks
  Arms: monotherapy

SUMMARY:
Hypothesis: Add-on therapy with oral montelukast (Mon) to inhaled budesonide (BUD) may achieve better control of cough caused by nonasthmatic eosinophilic bronchitis (NAEB) with faster reduction of airway eosinophilia.

Objective: To evaluate the efficacy of add-on therapy with Mon to inhaled corticosteroids (ICS) in the treatment of adult patients with chronic/subacute cough caused by NAEB diagnosed in outpatient setting. Primary endpoint：cough severity rated as cough visual analogue score (VAS)1 and eosinophil count in induced sputum during 4-week BUD monotherapy or Mon adjunct therapy.

DETAILED DESCRIPTION:
Subjects：63 newly-diagnosed, steroid-naïve adult patients with chronic or subacute cough caused by NAEB.

Grouping：ICS monotherapy (21 patients, BUD，400mcg mcg, twice daily+ placebo, 4 wks); Mon adjunct therapy (42 patients, Mon 10mg once daily + BUD 400mcg twice daily 4wks).

Protocol Day 1: In the respiratory specialist clinic, the diagnosis of NAEB is established following the 2006 ACCP guideline (sputum eosinophilia >3%, negative chest radiography, spirometry and bronchial provocation test). After briefing, eligible subjects who have given informed written consents, are to be randomly allocated to different treatment groups. Patients' demographical data, course and nature of cough, accompanying symptoms and upper respiratory comorbidities, skin prick test to common aeroallergens1, baseline cough VAS (0-100 mm) 1, spirometry and induced sputum cell counts, will be recorded by the managing physician in case record file (CRF). Pulmicort Turbuhaler (AstraZeneca, budesonide 100 mcg/dose X 200 doses) will be prescribed to each patient.

Day 2: Before initiation of treatment, at the Office for Clinical Trials, staff members will instruct the patients on correct usage of ICS, disperse Mon tablets or placebo as well as daily record cards, and explain how to record daily use of ICS and Mon, and adverse events. Once the treatment is initiated, oral steroids, other ICS, anti-histamines, beta-2 agonists and theophyllines will not be prescribed and used throughout the study period.

Day 8、15：Revisits: Patients' nature of cough, accompanying symptoms, cough VAS, induced sputum cell count will be reevaluated and recorded in CRF. Old daily record cards will be collected. New ones as well as Mon tablets or placebo will be given. Patients' skill of using ICS, compliance, systemic or local adverse events will be monitored.

Day 29： Revisit: Patients' nature of cough, accompanying symptoms, cough VAS, spirometry, bronchial provocation test, induced sputum cell count will be reevaluated and recorded in CRF. Old daily record cards will be collected. Patients' skill of using ICS, compliance, systemic or local adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult nonsmoking NAEB patients
* Without history of taking Mon, oral or inhaled corticosteroids, and
* Without bacterial or viral respiratory infections within 30 days prior to diagnosis of NAEB

Exclusion Criteria:

* Current smokers
* Pregnant or lactating women
* Known allergy to Mon, oral or inhaled corticosteroids
* Unable to use ICS following repeated instructions
* Complicated with unresectable malignancy or severe heart, lung, liver or kidney diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
cough severity rated as cough visual analogue score (VAS) | 4 weeks
eosinophil count in induced sputum | 4 weeks

SECONDARY OUTCOMES:
adverse reactions | 4 weeks
  any discomforts or untoward events observed during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Birring SS, Berry M, Brightling CE, Pavord ID. Eosinophilic bronchitis: clinical features, management and pathogenesis. Am J Respir Med. 2003;2(2):169-73. doi: 10.1007/BF03256647. PMID 14720015
- [Derived] Cai C, He MZ, Zhong SQ, Tang Y, Sun BQ, Chen QL, Zhong NS. Add-on montelukast vs double-dose budesonide in nonasthmatic eosinophilic bronchitis: a pilot study. Respir Med. 2012 Oct;106(10):1369-75. doi: 10.1016/j.rmed.2012.06.009. Epub 2012 Jul 21. PMID 22819521